CLINICAL TRIAL: NCT05277922
Title: A Phase 1, Open-label, Single-centre Study Investigating the Effect of C21 on Forearm Blood Flow in Healthy Male Subjects by Use of Strain-gauge Venous Occlusion Plethysmography
Brief Title: Effect of C21 on Forearm Blood Flow
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vicore Pharma AB (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: VP-C21-009
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Results first posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Study Vasodilatory Effects of C21
MeSH Terms: interventions — compound 21; Nitroprusside

STUDY DESIGN:
Intervention Model Description: Subjects will receive increasing doses of C21
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C21 combined (Experimental): 15 µg C21 (infusion rate 3 µg/min) 50 µg C21 (infusion rate 10 µg/min) 150 µg C21 (infusion rate 30 µg/min) 500 µg C21 (infusion rate 100 µg/min) 1000 µg C21 (infusion rate 200 µg/min)
  Interventions: Drug: C21
- Positive control (Experimental): 4 µg nitroprusside (infusion rate 0.8 µg/min) 8 µg nitroprusside (infusion rate 1.6 µg/min) 16 µg nitroprusside (infusion rate 3.2 µg/min)
  Interventions: Drug: Sodium Nitroprusside

INTERVENTIONS:
Drug: C21 — C21 in ascending doses of 15, 50, 150, 500 and 1000 µg
  Other Names: Compund 21
  Arms: C21 combined
Drug: Sodium Nitroprusside — Ascending doses of 4, 8 and 16 µg sodium nitroprusside Positive control
  Other Names: Nipruss
  Arms: Positive control

SUMMARY:
The purpose of this study is to assess the effect of C21 on forearm blood flow by use of strain-gauge venous occlusion plethysmography.

DETAILED DESCRIPTION:
Subject will be screened for eligibility. Eligible subjects will receive ascending doses of C21 (3, 10, 30, 100, and 200 µg/min through local intra-arterial infusions for 5 min/dose. Forearm blood flow measurements will be performed in both arms during the last 2 minutes of each dose.

Infusions of sodium nitroprusside will be performed as a positive control using the same methodology.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study and to comply with study requirements.
2. Healthy male subject aged 18-45 years
3. Body mass index ≥ 18.5 and ≤ 30.0 kg/m2.
4. Wlling to use condom or be vasectomised or practice sexual abstinence
5. Clinically normal medical history, physical findings, vital signs, ECG and laboratory values

Exclusion Criteria:

1. History of any clinically significant disease or disorder which may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. History of thrombotic disease, vascular disorder, or severe bleeding disease.
3. Poor brachial artery access.
4. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of baseline
5. Malignancy within the past 5 years with the exception of basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
6. Any planned major surgery within the duration of the study.
7. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody and human immunodeficiency virus (HIV).
8. Abnormal vital signs
9. Prolonged QT interval, cardiac arrhythmias or any clinically significant abnormalities in the resting ECG
10. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity or history of hypersensitivity to drugs with a similar chemical structure or class to the IMPs, including any of the excipients of the IMPs.
11. Regular use of any prescribed or non-prescribed medication including antacids, analgesics, herbal remedies, vitamins, and minerals
12. Regular use of non-steroidal anti-inflammatory drugs or acetylsalicylic acid
13. Vaccination within 1 week prior to dosing or plans to receive any vaccine during the study conduct.
14. Planned treatment or treatment with another investigational drug within 3 months
15. Current regular smokers or users of nicotine products.
16. History of alcohol abuse
17. Presence or history of drug abuse
18. Positive screen for drugs of abuse or alcohol at screening
19. History of, or current use of, anabolic steroids.
20. Inability to refrain from consuming caffeine-containing beverages during Day 1
21. Plasma donation within 1 month of screening or blood donation (or corresponding blood loss) during the 3 months prior to screening.
22. Investigator considers the subject unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Consultants AB, Uppsala, Uppsala Lân, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rein-Hedin E, Sjoberg F, Ganslandt C, Skoog J, Zachrisson H, Bengtsson T, Dalsgaard CJ. Utilizing venous occlusion plethysmography to assess vascular effects: A study with buloxibutid, an angiotensin II type 2 receptor agonist. Clin Transl Sci. 2024 Feb;17(2):e13735. doi: 10.1111/cts.13735. PMID 38344891

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 subjects were enrolled into the trial and all subjects received 5 ascending doses of C21 followed by 3 ascending doses of sodium nitroprusside as a positive control. Thus, the 5 subjects were reused for both C21 and sodium nitroprusside treatment.
Period: 15 µg C21
Arm/Group | C21 Combined | Positive Control
Started | 5 | 0
Completed | 5 | 0
Not Completed | 0 | 0
Period: 50 µg C21
Arm/Group | C21 Combined | Positive Control
Started | 5 | 0
Completed | 5 | 0
Not Completed | 0 | 0
Period: 150 µg C21
Arm/Group | C21 Combined | Positive Control
Started | 5 | 0
Completed | 5 | 0
Not Completed | 0 | 0
Period: 500 µg C21
Arm/Group | C21 Combined | Positive Control
Started | 5 | 0
Completed | 5 | 0
Not Completed | 0 | 0
Period: 1000 µg C21
Arm/Group | C21 Combined | Positive Control
Started | 5 | 0
Completed | 5 | 0
Not Completed | 0 | 0
Period: 4 µg Nitroprusside
Arm/Group | C21 Combined | Positive Control
Started | 0 | 5
Completed | 0 | 5
Not Completed | 0 | 0
Period: 8 µg Nitroprusside
Arm/Group | C21 Combined | Positive Control
Started | 0 | 5
Completed | 0 | 5
Not Completed | 0 | 0
Period: 16 µg Nitroprusside
Arm/Group | C21 Combined | Positive Control
Started | 0 | 5
Completed | 0 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | C21 Combined
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.0 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: cm] | 180.0 (7.1)
Weight [Mean (Standard Deviation); unit: kg] | 86.8 (9.1)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 26.8 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Forearm Blood Flow in Response to Increasing Intraarterial Doses of C21
Description: Percentage change from baseline in forearm blood flow (FBF) in response to increasing intraarterial doses of C21 (3, 10, 30, 100, and 200 μg/min)
Time Frame: 85 minutes
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Groups:
- C21 3 ug/Min: First dose of C21: 3 ug/min
- C21 10 ug/Min: Second dose of C21: 10 ug/min
- C21 30 ug/Min: Third dose of C21: 30 ug/min
- C21 100 ug/Min: Fourth dose of C21: 100 ug/min
- C21 200 ug/Min: Last dose of C21: 200 ug/min
Arm/Group | C21 3 ug/Min | C21 10 ug/Min | C21 30 ug/Min | C21 100 ug/Min | C21 200 ug/Min
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
percentage of change from baseline | 27.8 (24.3) | 17.2 (5.5) | 37.0 (26.6) | 28.5 (22.7) | 60.5 (38.3)

2. Secondary Outcome: Dose-response Curve of C21 on Forearm Blood Flow (FBF)
Description: Geometric mean forearm blood flow (mL/min) by increasing C21 dose (3, 10, 30, 100, and 200 μg/min)
Time Frame: 85 min
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | C21 3 ug/Min | C21 10 ug/Min | C21 30 ug/Min | C21 100 ug/Min | C21 200 ug/Min
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
mL/min | 2.594 (43.2) | 2.594 (32.4) | 3.231 (44.7) | 3.215 (38.1) | 3.907 (24.5)
Statistical Analysis 1: Comparison: C21 3 ug/Min vs C21 10 ug/Min; Test type: Superiority; Geometric mean ratio = 0.9999, 95% CI 2-sided [0.8313 to 1.2025]
Statistical Analysis 2: Comparison: C21 3 ug/Min vs C21 30 ug/Min; Test type: Superiority; Geometric mean ratio = 1.2454, 95% CI 2-sided [1.0355 to 1.4979]
Statistical Analysis 3: Comparison: C21 3 ug/Min vs C21 100 ug/Min; Test type: Superiority; Geometric mean ratio = 1.2392, 95% CI 2-sided [1.0304 to 1.4904]
Statistical Analysis 4: Comparison: C21 10 ug/Min vs C21 100 ug/Min; Test type: Superiority; Geometric mean ratio = 1.2394, 95% CI 2-sided [1.0305 to 1.4906]
Statistical Analysis 5: Comparison: C21 30 ug/Min vs C21 100 ug/Min; Test type: Superiority; Geometric mean ratio = 0.9950, 95% CI 2-sided [0.8273 to 1.1967]
Statistical Analysis 6: Comparison: C21 3 ug/Min vs C21 200 ug/Min; Test type: Superiority; Geometric mean ratio = 1.5058, 95% CI 2-sided [1.2520 to 1.8110]
Statistical Analysis 7: Comparison: C21 10 ug/Min vs C21 200 ug/Min; Test type: Superiority; Geometric mean ratio = 1.5060, 95% CI 2-sided [1.2522 to 1.8113]
Statistical Analysis 8: Comparison: C21 30 ug/Min vs C21 200 ug/Min; Test type: Superiority; Geometric mean ratio = 1.2091, 95% CI 2-sided [1.0053 to 1.4541]
Statistical Analysis 9: Comparison: C21 100 ug/Min vs C21 200 ug/Min; Test type: Superiority; Geometric mean ratio = 1.2151, 95% CI 2-sided [1.0103 to 1.4614]
Statistical Analysis 10: Comparison: C21 10 ug/Min vs C21 30 ug/Min; Test type: Superiority; Geometric mean ratio = 1.2456, 95% CI 2-sided [1.0357 to 1.4981]

3. Secondary Outcome: Percentage Change From Baseline in Forearm Blood Flow in Response to Increasing Intra-arterial Doses of Sodium Nitroprusside
Description: Percentage change from baseline in forearm blood flow in response to increasing intra-arterial doses of sodium nitroprusside (0.8, 1.6, and 3.2 μg/min)
Time Frame: 45 minutes
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Groups:
- Nipruss 0.8 ug/Min: First dose of nipruss 0.8 ug/min
- Nipruss 1.6 ug/Min: Second dose of nipruss 1.6 ug/min
- Nipruss 3.2 ug/Min: Last dose of nipruss 3.2 ug/min
Arm/Group | Nipruss 0.8 ug/Min | Nipruss 1.6 ug/Min | Nipruss 3.2 ug/Min
Number analyzed (Participants) | 5 | 5 | 5
percentage of change from baseline | 319.8 (186.0) | 229.5 (73.1) | 319.6 (141.4)

4. Secondary Outcome: Frequency of Adverse Events
Description: Total number of adverse events was counted
Time Frame: Day 1-7
Measure: Number; unit: Number of adverse events
Groups:
- C21 Group: Participants infused with increasing doses of C21
- Total: All participants (infused with C21 and nitroprusside)
Arm/Group | C21 Group | Total
Number analyzed (Participants) | 5 | 5
Number of adverse events | 3 | 3

5. Secondary Outcome: Number of Mild, Moderate, and Severe Adverse Events
Description: Number of mild, moderate, and severe adverse events was counted
Time Frame: Day 1-7
Measure: Number; unit: Number of events
Arm/Group | C21 Group | Total
Number analyzed (Participants) | 5 | 5
Number of events
  Number of mild AEs | 3 | 3
  Number of moderate Aes | 0 | 0
  Number of severe AEs | 0 | 0

6. Secondary Outcome: Number of Serious Adverse Events (SAEs)
Description: Number of serious adverse events (SAEs) was counted
Time Frame: Day 1-7
Measure: Number; unit: Number of SAEs
Arm/Group | C21 Group | Total
Number analyzed (Participants) | 5 | 5
Number of SAEs | 0 | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Sign Parameters
Description: Participants with Clinically significant changes from baseline (screening ) to the end of treatment in mean systolic blood pressure, diastolic blood pressure or pulse rate were counted
Time Frame: 5 hours
Measure: Count of Participants; unit: Participants
Arm/Group | C21 Group | Total
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Changes in ECG Parameters
Description: Participants with Clinically significant changes from baseline (screening ) to the end of treatment in mean values of the ECG parameters were counted
Time Frame: 5 hours
Measure: Count of Participants; unit: Participants
Arm/Group | C21 Group | Total
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Changes in Safety Laboratory Parameters
Description: Participants with Clinically significant changes from baseline (screening ) to the end of treatment (Day 1) in mean clinical chemistry, haematology or coagulation parameters were counted
Time Frame: 5 hours
Measure: Count of Participants; unit: Participants
Arm/Group | C21 Group | Total
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from trial start until end-of-trial contact (follow-up), 7 days after trial start
Description: Adverse events were recorded from trial start until end-of-trial contact (follow-up),
Arm/Group | C21 Group | Total
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/5 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C21 Group (N=5) | Total (N=5)
Infusion site bruising (General disorders) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/22/NCT05277922/Prot_SAP_000.pdf